CLINICAL TRIAL: NCT06527157
Title: PROspective ACcrual To Investigate reprOductive Cancers in womeN
Brief Title: Investigations of Reproductive Cancers in Women
Acronym: PROACTION:
Status: Recruiting | Type: Observational
Sponsor: PinkDx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PNK002
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Swab samples with DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign: sample collection from females with benign causes of AUB/PMB
- Malignant: sample collection from females with malignant causes of AUB/PMB

SUMMARY:
The goal of this study is to create a non-invasive diagnostic test to rule out gynecological cancer in females aged 45 and older with abnormal uterine or postmenopausal bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent form indicating that the subject has been informed of all pertinent aspects of the study.
2. Willing and able to comply with scheduled visits, study plan, and other procedures.
3. Expected to be available for the duration of the study and can be contacted by telephone during study participation.
4. Females aged 45 and older (with roughly 80% of enrolled subjects over the age of 50).
5. Presence of uterus.
6. AUB or PMB being worked up to diagnose the cause of the bleeding

Exclusion Criteria:

1. Investigator site staff members directly involved in the conduct of the study and their family members or subjects who are PinkDx, Inc. employees or their family members.
2. Other medical or psychiatric conditions that would increase the risk of study participation in the judgement of the Investigator.
3. Women who have had a hysterectomy.
4. Women with a known history of endometrial cancer or uterine sarcoma.
5. Women who have received prior treatment for endometrial cancer.
6. Inability or unwillingness to sign informed consent.
7. Clinical suspicion of pregnancy.
8. Women who have used a tampon within 7 days of sample collection.

Ages: 45 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Females 45 years and older seeking medical attention for abnormal uterine or postmenopausal bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 12 months
  ability to detect cancer

SECONDARY OUTCOMES:
Specificity | 12 months
  ability to identify benign cases

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Mariani, MD, Principal Investigator — Mayo Clinic
Locations (16):
- United States (16):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Sutter Health, Redwood City, California
  - Advent Health Orlando, Orlando, Florida
  - Ob-Gyne Associates of Lake Forest, Ltd, Lake Forest, Illinois
  - Indiana University, Eskenazi Health, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University, New York, New York
  - Summa Health, Akron, Ohio
  - The Ohio State University, Columbus, Ohio
  - Avera Research Institute, Sioux Falls, South Dakota
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Houston Methodist, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No